CLINICAL TRIAL: NCT05149716
Title: Taurine as a Possible Anti-aging Therapy? A Controlled Clinical Trial on Taurine Antioxidant Activity in Women Aged 55 to 70 Years
Brief Title: Taurine as a Possible Anti-aging Therapy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Taurine_aging
Record Dates: First submitted 2021-11-19; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Oxidative Stress
Keywords: Aging; Oxidative Stress; Taurine; Nutritional Supplementation; Therapeutic Strategy
MeSH Terms: interventions — Taurine

STUDY DESIGN:
Intervention Model Description: Double-blind placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Supplement capsule packages were labeled as "Supplement A" and "Supplement B" and the nutrient (taurine or placebo- starch) was revealed after the end of the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taurine supplementation (Experimental): Taurine supplementation composed of capsules of taurine powder. Dosage: 1.5 gram/day Frequency: 1 time/day Duration: 16 weeks
  Interventions: Dietary Supplement: Taurine
- Placebo supplementation (Placebo Comparator): Placebo supplementation composed of capsules of starch powder. Dosage: 1.5 gram/day Frequency: 1 time/day Duration: 16 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Taurine — Taurine supplementation in capsules of 500 grams of taurine powder, total dosage: 1.5 gram/day
  Other Names: Taurine supplementation in capsules of 500 grams of taurine powder, total dosage: 1.5 grams/day
  Arms: Taurine supplementation
Dietary Supplement: Placebo — Placebo supplementation in capsules of 500 grams of starch powder, total dosage: 1.5 gram/day
  Arms: Placebo supplementation

SUMMARY:
Among the strategies that can improve the body's ability to counteract oxidative stress, the use of nutritional antioxidants has been investigated. Taurine is a "semi-essential" amino acid, also called a nitrogen compound, which has been used as an effective antioxidant due to its ability to neutralize hypochlorous acid, an extremely toxic oxidant produced by leukocytes in the inflammatory process in humans.

DETAILED DESCRIPTION:
Objective: To evaluate the oxidative parameters of women aged 55 to 70 years after 16 weeks of taurine supplementation.

Methods: Twenty-four women age 55 to 70 will be randomly assigned to two groups: control group (GC), supplemented with placebo (1.5 g of starch); and taurine group (GTAU), supplemented with taurine (1.5 g), for 16 weeks. Anthropometry, functional capacity test, taurine, and levels of oxidative stress markers will be determined in pre and post intervention plasma samples. Food consumption will be assessed before, during, and after the intervention. The results will be analyzed by an ANOVA two-way repeated measures mixed model, with the Sidak post hoc (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Had being aged 55-70 years;
* Female;
* Post-menopausal;
* Sedentary (not practicing physical exercise for at least 6 months).

Exclusion Criteria:

* Chronic kidney diseases;
* Infectious contagious diseases;
* Coronary heart disease;
* Smokers
* Alcoholics.

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood oxidative stress marker measurement - Superoxide Dismutase (SOD). | sixteen weeks
  The superoxide dismutase (SOD) activity in erythrocytes was evaluated by the spectrophotometric method, and were calculated at 16 weeks in comparision to the baseline.
Change from baseline in blood oxidative stress marker measurement - Glutathione reductase (GR). | sixteen weeks
  Glutathione reductase (GR) activity was determined by the spectrophotometric method at 37 ºC/340nm after the oxidation of NADPH in the presence of oxidized glutathione, and were calculated at 16 weeks in comparision to the baseline.
Change from baseline in blood oxidative stress marker measurement - Malondialdehyde (MDA). | sixteen weeks
  The malondialdehyde (MDA) were calculated at 16 weeks in comparision to the baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C Freitas, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Escola de Educação Física e Esporte de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schaffer S, Kim HW. Effects and Mechanisms of Taurine as a Therapeutic Agent. Biomol Ther (Seoul). 2018 May 1;26(3):225-241. doi: 10.4062/biomolther.2017.251. PMID 29631391
- [Background] Tadolini B, Pintus G, Pinna GG, Bennardini F, Franconi F. Effects of taurine and hypotaurine on lipid peroxidation. Biochem Biophys Res Commun. 1995 Aug 24;213(3):820-6. doi: 10.1006/bbrc.1995.2203. PMID 7654243
- [Background] Oliveira MW, Minotto JB, de Oliveira MR, Zanotto-Filho A, Behr GA, Rocha RF, Moreira JC, Klamt F. Scavenging and antioxidant potential of physiological taurine concentrations against different reactive oxygen/nitrogen species. Pharmacol Rep. 2010 Jan-Feb;62(1):185-93. doi: 10.1016/s1734-1140(10)70256-5. PMID 20360629
- [Background] Lourenco R, Camilo ME. Taurine: a conditionally essential amino acid in humans? An overview in health and disease. Nutr Hosp. 2002 Nov-Dec;17(6):262-70. PMID 12514918
- [Background] Sun Jang J, Piao S, Cha YN, Kim C. Taurine Chloramine Activates Nrf2, Increases HO-1 Expression and Protects Cells from Death Caused by Hydrogen Peroxide. J Clin Biochem Nutr. 2009 Jul;45(1):37-43. doi: 10.3164/jcbn.08-262. Epub 2009 Jun 30. PMID 19590705
- [Background] Rosa FT, Freitas EC, Deminice R, Jordao AA, Marchini JS. Oxidative stress and inflammation in obesity after taurine supplementation: a double-blind, placebo-controlled study. Eur J Nutr. 2014 Apr;53(3):823-30. doi: 10.1007/s00394-013-0586-7. Epub 2013 Sep 25. PMID 24065043
- [Background] De Carvalho FG, Galan BSM, Santos PC, Pritchett K, Pfrimer K, Ferriolli E, Papoti M, Marchini JS, de Freitas EC. Taurine: A Potential Ergogenic Aid for Preventing Muscle Damage and Protein Catabolism and Decreasing Oxidative Stress Produced by Endurance Exercise. Front Physiol. 2017 Sep 20;8:710. doi: 10.3389/fphys.2017.00710. eCollection 2017. PMID 28979213
- [Background] Chupel MU, Minuzzi LG, Furtado GE, Santos ML, Ferreira JP, Filaire E, Teixeira AM. Taurine supplementation reduces myeloperoxidase and matrix-metalloproteinase-9 levels and improves the effects of exercise in cognition and physical fitness in older women. Amino Acids. 2021 Mar;53(3):333-345. doi: 10.1007/s00726-021-02952-6. Epub 2021 Feb 13. PMID 33586039
- [Result] Marcinkiewicz J, Kontny E. Taurine and inflammatory diseases. Amino Acids. 2014 Jan;46(1):7-20. doi: 10.1007/s00726-012-1361-4. Epub 2012 Jul 19. PMID 22810731